CLINICAL TRIAL: NCT01538225
Title: Neurophysiologic Study on Effects of Sativex® on Spasticity in Progressive Multiple Sclerosis
Brief Title: Neurophysiological Study of Sativex in Multiple Sclerosis (MS) Spasticity
Acronym: NS-MSS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: M/SATIVX/01; 2011-002258-30 (EudraCT Number)
Record Dates: First submitted 2012-02-20; First posted 2012-02-24 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Multiple Sclerosis
Keywords: Spasticity
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- first sativex, second placebo (Experimental): 2 weeks first titration period (as per approved SmPC), a 2-week first treatment period (Sativex), a 2-week washout, a cross-over followed by another 2 weeks titration period (as per SmPC), followed by a second 2-week period treatment (placebo)
  Interventions: Drug: Sativex®; Drug: Placebo
- first placebo, second sativex (Experimental): 2 weeks first titration period (as per approved SmPC), a 2-week first treatment period (placebo), a 2-week washout, a cross-over followed by another 2 weeks titration period (as per SmPC), followed by a second 2-week period treatment (Sativex)
  Interventions: Drug: Sativex®; Drug: Placebo

INTERVENTIONS:
Drug: Sativex® — THC:CBD 1:1 ratio oromucosal spray. A titration period is required to reach optimal dose. The number and timing of sprays may vary between patients.
  Duration: 2 weeks
Drug: Placebo — Placebo
  Same frequency and dosage form as Sativex.
  Duration: 2 weeks

SUMMARY:
Aim of this randomized, double-blind, placebo-controlled, cross-over study is to investigate cannabinoid-induced changes in neurophysiological parameters in a group of 40 patients with secondary or primary progressive Multiple Sclerosis (MS).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or above
* Willing and able to comply with the protocol for the duration of the study
* Diagnosis of Secondary-Progressive or Primary-Progressive MS from at least 12 months
* Relapse free from at least 3 months before screening visit
* Lower limb spasticity
* EDSS from > 3.0 and < 6.5
* Moderate to severe spasticity due to MS from at least 6 months and with stable drug treatment not able to relieve symptoms as a whole, deserving a specific add-on treatment
* Immunomodulatory or immunosuppressant therapies not modified during the study and 6 months before starting the study
* Stable doses of anti-spasticity agents from at least 2 months prior to screening visit
* Have given written informed consent

Exclusion Criteria:

* Any concomitant disease that may cause spasticity or that could interfere with subject's spasticity
* Botulinum Toxin injection for spasticity in the 4 months prior to screening visit
* Any known or suspected history of psychotic illness, alcohol or substance abuse, epilepsy, hypersensitivity to cannabinoids
* Significant cardiac, renal or hepatic disease
* Female subjects of child bearing potentials and male subjects whose partner is child bearing potential, unless willing to ensure that they or their partner use contraception during the study
* Female subjects who is pregnant lactating or planning pregnancy during the course of the study and for three months thereafter
* Sativex® SmPC contraindications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
H/M reflex ratio | week 0, 4
  To evaluate differences in the H/M ratio scores within subjects affected by progressive MS at baseline and week 4.

SECONDARY OUTCOMES:
Neurophysiology ·H/M ratio ·Transcranial Magnetic Stimulation a) MEP Motor threshold, upper limb b) MEPs amplitudes c) Intracortical facilitation/inhibition (ICI/ICF), upper limb | week 0, 4, 6 and 10
  Neurophysiology
  * H/M ratio: To evaluate differences in the H/M ratio scores within subjects affected by progressive MS at weeks 6 and 10
  * Transcranial Magnetic Stimulation
    1. Motor threshold to obtain MEPs to the upper limb (time 0-4; 6-10 weeks);
    2. MEPs amplitudes at 15% above motor threshold, measured as MEP/M ratio to APB (abductor pollicis brevis) and abductor of hallucis, in which M is the compound muscle potential in response to peripheral stimulation (time 0-4; 6-10 weeks);
    3. Intracortical facilitation/inhibition (ICI/ICF) to the upper limb (time 0-4; 6-10 weeks);
Adverse Events recording | week 0, 4, 6 and 10
Spasticity: ·0-10 11-point numerical spasticity rating scale (NRS) ·Mean modified Ashworth scale (MAS) | week 0, 4, 6, 10
  Mean spasticity score recorded using a 0-10 11-point numerical spasticity rating scale (NRS) at baseline (pre-treatment) and week 4, 6 and 10
  · Mean modified Ashworth (MAS) score at baseline (pre-treatment), week 4, 6, 10
Function: ·Timed 25 feet and 10 meters walk ·Hand dexterity measured with 9-HPT | week 0, 4, 6, 10
  Function:
  * Mean Timed 25 feet and 10 meters walk recorded at baseline (pre-treatment) and week 4, 6, 10
  * Mean Hand dexterity measured with 9-HPT recorded at baseline (pre-treatment) and week 4, 6, 10
Other MS Symptoms: ·Sleep Quality NRS ·Pain NRS and Spasm frequency ·Fatigue Severity Scale (FSS) | week 0, 4, 6, 10
  Other MS Symptoms:
  * Mean Sleep Quality NRS recorded at baseline (pre-treatment) and week 4, 6, 10
  * Pain NRS and Spasm frequency recorded at baseline (pre-treatment) and week 4, 6, 10
  * Fatigue measured with the Fatigue Severity Scale (FSS) recorded at baseline (pre-treatment) and week 4, 6, 10

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Comi, Prof, Principal Investigator — Institute of Experimental Neurology (Milan, Italy)
Locations (1):
- Institute of Experimental Neurology, Milan, Italy